CLINICAL TRIAL: NCT02972515
Title: Mobile Application for Guided Imagery to Address Smoking, Diet and Physical Activity
Acronym: Imagery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: West Virginia University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21CA174639 (NIH); 1R21CA174639 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2016-11

CONDITIONS: Smoking Cessation
Keywords: Smoking; Smoking cessation; Multiple behaviors; mHealth; Mobile Application
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- See Me Smoke-Free (Experimental): Participants received access to the See Me Smoke-Free mobile application (app) delivered via smart phone, and were asked to use the app "most days" for 30 days post-enrollment. The app contained five guided imagery audio files (Introduction to Guided Imagery, Be Smoke Free, Eat Well, Get Active, and Feel Fantastic), a tracking calendar, awards, resources, reminders, and tips and techniques.
  Interventions: Behavioral: See Me Smoke-Free; Device: Smart phone

INTERVENTIONS:
Behavioral: See Me Smoke-Free — See Me Smoke-Free is a multi-behavioral mobile application focusing on increasing smoking cessation, healthy eating, and moderate to intense physical activity. The app tracks the participant's quit date, and eating/physical activity goals. Participants have access to guided imagery audio files that they are instructed to listen to every day for at least 30 days. Participants can earn awards for meeting the study goals.
Device: Smart phone — See Me Smoke-Free mHealth app delivered via a smart phone

SUMMARY:
Tobacco use among women now approaches that of men, with approximately 27 million women smokers in the United States alone. Women report greater difficulties quitting smoking and are more likely to relapse than men. In addition, tobacco use co-varies with poor dietary practices and lack of physical activity, with 92% of smokers reporting at least one other health risk factor. Concerns surrounding weight gain, negative body image, and low self-efficacy, may be key factors affecting smoking cessation among weight-concerned women smokers. Guided imagery has been successfully employed in separate lines of inquiry to address physical activity, diet and smoking cessation. However, guided imagery has not been employed to target weight concerned women who smoke or to simultaneously target smoking, diet, and exercise behavior in a single intervention. The proposed study would be the first of its kind to create a theory-based, guided imagery intervention to assist weight-concerned women smokers to quit. The use of a mobile app offers an innovative approach to addressing the multiple behaviors involved in smoking cessation efforts of weight-concerned women, and has the potential to reach large numbers of women smokers. The project aims to develop and test the feasibility of a mobile health application using guided imagery in order to increase smoking cessation among a population of weight-concerned women smokers.

DETAILED DESCRIPTION:
SPECIFIC AIMS Tobacco use among women now approaches that of men, with approximately 27 million women smokers in the United States alone. Lung cancer is the leading cause of cancer death among women, and more than 180,000 women die of other illnesses linked to smoking annually. Women report greater difficulties quitting smoking and are more likely to relapse than men. In addition, tobacco use co-varies with poor dietary practices and lack of physical activity, with 92% of smokers reporting at least one other health risk factor. The presence of multiple behavioral risk factors greatly increases the risk of developing many acute and chronic conditions.

Concerns about weight gain, negative body image, and lack of self-efficacy may be key factors affecting smoking, diet, and exercise behavior of women. Women smokers are less satisfied with their bodies, have lower self-esteem, and are more concerned about becoming overweight than non-smokers. Approximately 50% of women smokers report that concerns about body weight are reasons they do not quit. Research indicates that women report lower self-efficacy in quitting than men, especially women concerned about controlling their weight. These findings suggest that targeting weight concerns, body image, and self-efficacy to quit with weight-concerned women who smoke may be an effective intervention strategy. Recent studies suggest that a multi-behavioral approach, including diet and physical activity, may be more effective at helping weight-concerned smokers to quit.

One cognitive approach, guided imagery, has been successfully employed in separate lines of inquiry to address body image concerns and self-efficacy in our three target behaviors-exercise, diet and smoking cessation. However, guided imagery has not been employed to target weight concerned women who smoke or to simultaneously target smoking, diet, and exercise behavior in a single intervention. The proposed study would be the first of its kind to create a theory-based, guided imagery intervention to assist weight-concerned women smokers to quit.

While imagery is an effective therapeutic tool for behavior change, the mode of delivery has generally been in-person, limiting the dissemination of guided imagery-based interventions to large populations. Mobile health applications (mobile apps) delivered via smart phones offer a unique channel through which to distribute imagery-based interventions. Mobile apps may enhance the use of guided imagery through the use of audio files. The app may allow guided imagery scripts to be tailored by the user, and flexibly administered at varying times (e.g., during nicotine cravings). This approach could be especially useful for women, who are more likely than men to use the Internet to obtain health information. The use of a mobile app offers an innovative approach to addressing the multiple behaviors involved in smoking cessation efforts of weight-concerned women, and has the potential to reach large numbers of women smokers. If successful, a mobile application for guided imagery could be used to address other health behaviors as well. The present project aims to develop and test the feasibility of a mobile health application using guided imagery in order to increase smoking cessation among weight-concerned women smokers.

The Specific Aims for this study are to:

Aim 1. Develop guided imagery content, user interface, and resources to reduce weight concern, and increase body image and self-efficacy for behavior change among weight-concerned women smokers. Scripts incorporating imagery across these domains will be developed specifically for smoking cessation, eating a healthy diet and engaging in physical activity. The investigators will develop initial content and user interface ideas based on experience in using guided imagery for increasing physical activity, and using technology to assist tobacco cessation and healthy eating. Ten focus group participants (weight-concerned women smokers who own a smart phone, representing various racial/ethnic groups) will provide feedback on content, potential tailoring of content by race/ethnicity, functions, and design, which will inform development of the mobile app.

Aim 2. Program a prototype of the app that contains all the necessary elements of text, graphics, multimedia and interactive features. Users will be able to customize certain elements of the application, and be required to provide input in response to app prompts. The investigators will conduct usability testing, observing 10 participants using "think aloud" procedures as they interact with the app, to ensure that it is fully functional and easy to use.

Aim 3. Evaluate the feasibility, acceptability, and preliminary efficacy of the app with 50 weight-concerned women smokers. The primary outcome will be self-reported tobacco abstinence at 3 months post-enrollment. The investigators will also measure: dietary intake; level of physical activity; body image; self-efficacy; cravings; and participants' use of the app, including the imagery scripts, diary, and resource links.

The potential impact of this proposed intervention is great, because it addresses behavioral risk factors that can be applied to populations beyond smokers. This proposal is significant because it intervenes with women smokers; innovative, in that it uses guided imagery to change lifestyle behaviors important for the prevention of chronic diseases, and, technology to maximize dissemination potential. The proposed investigation takes a theory-based approach, builds on the considerable track records of the investigators, and will be conducted in an environment highly suited for this study. Results of this study will be used to prepare for a future randomized controlled trial to test the efficacy and cost-effectiveness of a multi-behavioral, guided imagery mobile health application versus a single smoking cessation imagery mobile health application.

ELIGIBILITY:
Inclusion Criteria include the following:

* Must be female
* Report smoking in the past 30 days
* Use an Android cell phone
* Have a valid email address
* Have a valid phone number
* Speak English

Exclusion Criteria including the following:

* Male
* Not a current smoker
* Do not use an Android cell phone
* Do not have a valid email address
* Do not have a valid phone number
* Do not speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Gordon, PhD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giacobbi P Jr, Hingle M, Johnson T, Cunningham JK, Armin J, Gordon JS. See Me Smoke-Free: Protocol for a Research Study to Develop and Test the Feasibility of an mHealth App for Women to Address Smoking, Diet, and Physical Activity. JMIR Res Protoc. 2016 Jan 21;5(1):e12. doi: 10.2196/resprot.5126. PMID 26795257
- [Background] Armin J, Johnson T, Hingle M, Giacobbi P Jr, Gordon JS. Development of a Multi-Behavioral mHealth App for Women Smokers. J Health Commun. 2017 Feb;22(2):153-162. doi: 10.1080/10810730.2016.1256454. Epub 2017 Jan 25. PMID 28121240

RESULTS

PARTICIPANT FLOW:
Groups:
- See Me Smoke-Free: Participants received access to the See Me Smoke-Free mobile application (app), and were asked to use the app "most days" for 30 days post-enrollment. The app contained five guided imagery audio files (Introduction to Guided Imagery, Be Smoke Free, Eat Well, Get Active, and Feel Fantastic), a tracking calendar, awards, resources, reminders, and tips and techniques.
  See Me Smoke-Free: See Me Smoke-Free is a multi-behavioral mobile application focusing on increasing smoking cessation, healthy eating, and moderate to intense physical activity. The app tracks the participant's quit date, and eating/physical activity goals. Participants have access to guided imagery audio files that they are instructed to listen to every day for at least 30 days. Participants can earn awards for meeting the study goals.
  Smart phone: See Me Smoke-Free mHealth app delivered via a smart phone
Period: Overall Study
Arm/Group | See Me Smoke-Free
Started | 166
Completed | 88
Not Completed | 78
Not completed — Lost to Follow-up | 78

BASELINE CHARACTERISTICS:
Population: Data reported for 73 participants who completed the feasibility trial. These data do not include participants from the formative phase of the study or those lost to follow-up.
Arm/Group | See Me Smoke-Free
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 53
  More than one race | 3
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 73
Smoked last 30 days [Count of Participants; unit: Participants] | 73
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per Day] | 16.0 (13.2)
Weight [Mean (Standard Deviation); unit: pounds] | 169.8 (43.0)
Frequency of fruit intake [Mean (Standard Deviation); unit: servings of fruit per day] | 3.70 (1.91)
Minutes of Exercise per Day [Mean (Standard Deviation); unit: Minutes of exercise per day] | 25.48 (23.75)
Use of any guided imagery [Mean (Standard Deviation); unit: minutes of any guided imagery daily] | 1.77 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Smoking Abstinence
Description: Self-reported smoking abstinence will be collected via online questionnaire at 3-months post-enrollment.
Time Frame: 3 months
Population: 63 feasibility participants with both baseline and 3-month data.
Measure: Count of Participants; unit: Participants
Arm/Group | See Me Smoke-Free
Number analyzed (Participants) | 63
Participants | 30

2. Secondary Outcome: Weekly Minutes of Exercise
Description: Self-reported level of moderate to strenuous physical activity will be collected via online questionnaire at 3-months post-enrollment.
Time Frame: 3 months
Population: Data analyzed on 60 feasibility participants with both baseline and 3-month data.
Measure: Mean (Standard Deviation); unit: minutes of exercise per week
Arm/Group | See Me Smoke-Free
Number analyzed (Participants) | 60
minutes of exercise per week | 269 (161)

3. Secondary Outcome: Servings of Fruit Per Day
Description: Self-reported consumption of servings of fruits per day will be collected via online questionnaire at 3-months post-enrollment.
Time Frame: 3 months
Population: 62 feasibility participants with data from both baseline and follow-up
Measure: Mean (Standard Deviation); unit: servings of fruit per day
Arm/Group | See Me Smoke-Free
Number analyzed (Participants) | 62
servings of fruit per day | 5.0 (202)

4. Secondary Outcome: Minutes of Guided Imagery Use Per Day
Description: Interaction with the mHealth app will be measured automatically and unobtrusively by the app on an on-going basis. The app will collect the number of minutes per day that the guided imagery audio files are listened to.
Time Frame: Collected throughout each day for up to 90 days
Population: 62 feasibility participant with both baseline and 3-month data.
Measure: Mean (Standard Deviation); unit: minutes of guided imagery user per day
Arm/Group | See Me Smoke-Free
Number analyzed (Participants) | 62
minutes of guided imagery user per day | 2.7 (1.2)

ADVERSE EVENTS:
Time Frame: 1 year
Description: This was an exempt study. There was no risk of mortality or serious adverse events as a result of this behavioral smoking cessation intervention.
Arm/Group | See Me Smoke-Free
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73
Other Adverse Events (participants affected / at risk) | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No